CLINICAL TRIAL: NCT00258479
Title: Modafinil and Nicotine in Adolescents: Phase I Trial
Brief Title: Safety of Combining Modafinil and Nicotine Replacement Therapy in Treating Nicotine Dependent Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Martin, MD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Catherine Martin, MD, Princial Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-15413; R03DA015413 (NIH); DPMCDA
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2012-03

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine Dependence; Nicotine Use Disorder; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Modafinil (Experimental)
  Interventions: Drug: ModafinilNicotine Replacement Therapy; Drug: Modafinil
- Placebo (Placebo Comparator)
  Interventions: Drug: ModafinilNicotine Replacement Therapy; Drug: Modafinil
- Nicotine Replacement Therapy (No Intervention): The effects of nicotine replacement therapy will be investigated - alone and in combination with modafinil - on nicotine withdrawal in nicotine-dependent adolescents.

INTERVENTIONS:
Drug: ModafinilNicotine Replacement Therapy — A dose escalation design includes eight dose conditions across a 12-day study (nicotine low-high, modafinil low-high and 4 combinations). After day 1 placebo dose, placebo sessions occur in random order during low dose, high dose, and dose-combination testing. Modafinil and nicotine are tested alone with subjects exposed to low active doses prior to higher doses. Dose interactions will be determined with low doses tested in combination followed by low-high dose combinations then high-high dose combination. Doses are administered under double-blind, double dummy procedures. A nicotine patch (0, 7 or 14 mg doses) is applied at 7 am. Modafinil doses are prepared in size 00 opaque capsules. The modafinil dose (0, 100, 200 mg) is administered at 5 PM.
  Other Names: Provigil
  Arms: Modafinil; Placebo
Drug: Modafinil — See Modafinil Intervention Description above.
  Other Names: Provigil
  Arms: Modafinil; Placebo

SUMMARY:
Nicotine is one of the most widely abused substances in the United States. Nicotine replacement therapy (NRT) is currently an effective treatment for nicotine dependence; however, even with NRT most people fail at quitting smoking after their first attempt. Modafinil is a promising drug that may be useful in treating nicotine dependent individuals. The purpose of this study is to evaluate the safety of the combination of modafinil and NRT in treating nicotine dependent adolescent smokers.

DETAILED DESCRIPTION:
NRT is a critical part of treating nicotine withdrawal symptoms, such as cravings, sleeplessness, poor concentration, and anxiety. The addition of modafinil, a promising pharmacologic agent, may enhance the effectiveness of NRT by further reducing inattention and depressed mood. The purpose of this study is to examine the safety of using both modafinil and NRT in treating nicotine dependent adolescents. In addition, this study will examine the effects of modafinil and NRT, alone and in combination, on alleviating symptoms of inattention and depressed mood.

Participants in this 12-day dose escalation study will be tested under eight different dose conditions. Modafinil and NRT will first be tested alone; participants will be exposed to low doses prior to higher doses of medication. Various modafinil-NRT dose combinations will then be tested. Modafinil will be administered at 5 p.m. each day, and NRT will be self-administered at the start of each day in which a participant must complete lab tests. The following measures will be obtained at study visits occurring before and after the various modafinil-NRT dose combinations: nicotine withdrawal symptoms, medication side effects, activity level, cardiovascular response, and profile of mood states (POMS).

ELIGIBILITY:
Inclusion Criteria:

* Smokes 10 or more cigarettes per day

Exclusion Criteria:

* Current use of any medication for a psychiatric disorder
* Positive drug screen test
* Uses smokeless tobacco

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2003-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety of combination drug treatment and physiological response; measured after treatment with each dose combination | laboratory session

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Martin, PhD, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States